CLINICAL TRIAL: NCT01262911
Title: A Phase I Study to Evaluate a Single Oral Dose of SRT2379 on the Endotoxin Induced Inflammatory Response in Healthy Male Subjects
Brief Title: Effect of SRT2379 on Endotoxin-Induced Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 115083
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 g SRT2379 (Active Comparator): Single dose of 1.0g of SRT2379
  Interventions: Drug: SRT2379
- 1.0 g Placebo (Placebo Comparator): Single dose of 1.0g of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRT2379 — SRT2379 will be supplied as hard gelatin capsules, with each containing 250mg.
  Arms: 1.0 g SRT2379
Drug: Placebo — Matching placebo will be supplied as hard gelatin capsules, with each containing an appropriate amount of placebo.
  Arms: 1.0 g Placebo

SUMMARY:
SRT2379 is a potent small molecule activator of SIRT1 that has been found to inhibit systemic inflammation induced by intravenous injection of lipopolysaccharide (LPS) in mice. The objective of this study is to test if SRT2379 may be a novel compound for the treatment of inflammatory disorders in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination and laboratory tests carried out within 21 days prior to dosing.
* Male between 18 and 35 years of age inclusive, at the time of signing the informed consent
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Chemistry panel, including renal and liver functions tests, without any clinically relevant abnormality
* Subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 7 days following the dose of study drug

Exclusion Criteria:

* Subject has had a major illness in the past 3 months or any significant chronic medical illness that the investigator would deem unfavorable for enrollment including inflammatory diseases
* Subjects with a history of any type of malignancy with the exception of successfully treated basal cell cancer of the skin
* Subject has a past or current gastrointestinal disease which may influence drug absorption
* The subject has a known positive test for hepatitis C antibody, hepatitis B surface antigen or HIV
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subject has a history, within three years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, THC) or a positive drug results at the Screening visit
* History of alcoholism and/or is drinking more than 3 drinks per day. Alcoholism is defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* The subject has participated in a clinical trial and has received an investigational product within three months of the dosing in the current study
* Use of prescription or non-prescription drugs, and herbal and dietary supplements within 7 days unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* Subject has difficultly in donating blood or accessibility of a vein in left or right arm
* Subject has donated more than 350 mL of blood in last 3 months
* Subject uses tobacco products
* Any clinically relevant abnormality noted on the 12-lead ECG as judged by the investigator or an average QTcB or QTcF > 450 msec
* Any other issue that, in the opinion of the Principal Investigator, would could be harmful to the subject or compromise interpretation of the data
* Prior participation in a trial where the subject received IV LPS

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02-17 (Actual); Primary Completion 2011-04-26 (Actual); Study Completion 2011-04-26 (Actual)

PRIMARY OUTCOMES:
To determine if a single dose of SRT2379 attenuates the inflammatory response in normal healthy male subjects after exposure to low-dose endotoxin (LPS). | 24 hours

SECONDARY OUTCOMES:
To determine PK of SRT2379 in normal healthy male subjects exposed to low-dose endotoxin (LPS). | 24 hours
To determine the safety profile of SRT2379 in healthy male subjects exposed to low-dose endotoxin (LPS). | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115083 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115083?search=study&study_ids=115083#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115083 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register